CLINICAL TRIAL: NCT07260526
Title: Response-adapted Total Neoadjuvant Therapy Guided by Induction Chemotherapy in Early- and Intermediate-risk Low Rectal Cancer for Implementation of a Watch-and-wait Strategy
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Director of Colorectal Surgery, Clinical Professor, West China Hospital
Other Study IDs: WCH20250924
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; total neoadjuvant therapy; watch-and-wait strategy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ITNT group: Patients who achieve a good response after total neoadjuvant therapy and receive organ preservation strategy

SUMMARY:
This study investigates the feasibility of an organ-preserving "watch-and-wait" strategy in patients with mid-to-low rectal cancer who achieve a good response after total neoadjuvant therapy (TNT). By retrospectively and prospectively analyzing patients who complete TNT following effective induction chemotherapy, the study aims to assess organ preservation rates and evaluate whether non-surgical management can provide comparable oncologic outcomes to radical surgery while improving functional recovery and quality of life.

DETAILED DESCRIPTION:
With the evolution of rectal cancer treatment concepts, achieving optimal oncologic outcomes while preserving organ function and improving patients' quality of life has become a major goal in the management of low rectal cancer. Multiple studies have reported that for patients who achieve a clinical complete response (cCR) after total neoadjuvant therapy (TNT), a watch-and-wait (organ preservation) strategy-with close follow-up and salvage surgery when necessary-yields 5-year disease-free survival (DFS) and overall survival (OS) rates comparable to those of patients who undergo radical surgery and achieve a pathological complete response (pCR). Moreover, compared with total mesorectal excision (TME), patients managed with a watch-and-wait approach demonstrate significantly better physical, cognitive, role, and social-emotional functioning, along with lower incidences of bowel, sexual, and urinary dysfunction.

This study aims to retrospectively and prospectively include patients with mid-to-low rectal cancer who respond well to induction chemotherapy and subsequently complete TNT, in order to observe the organ preservation rate after TNT and to preliminarily evaluate the feasibility of this treatment approach within a watch-and-wait strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years; no restriction on sex.
* Histologically confirmed rectal adenocarcinoma with immunohistochemistry and/or genetic testing showing pMMR/MSS status.
* Tumor characteristics assessed by chest-abdominal CT, rectal ultrasound, and MRI meeting all of the following criteria:

  1. The lower edge of the tumor is ≤5 cm from the anal verge as measured by digital rectal examination or MRI;
  2. Clinical stage cT1-3abN0-1M0 (for cT1N0, patients suitable for endoscopic resection are excluded);
  3. MRF (-) (>1 mm), EMVI (±);
  4. Negative lateral lymph nodes and <7 mm in size;
  5. Maximum tumor length ≤5 cm;
  6. Tumor circumference involvement ≤2/3.
* After receiving at least two cycles of induction chemotherapy with the XELOX regimen, MRI assessment shows treatment response (tumor length reduced by ≥30% compared with baseline).
* Completion of total neoadjuvant therapy (TNT), including long-course chemoradiotherapy and consolidation chemotherapy (radiotherapy: 25-28 fractions; chemotherapy: 6-8 cycles).
* (For the prospective cohort) Provision of written informed consent for participation in this observational study.

Exclusion Criteria:

* Patients with a history of, or concurrent, other malignant tumors (except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix);
* Patients with severely incomplete clinical data that preclude effective evaluation;
* (For the prospective cohort) Patients who refuse to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mid-to-low rectal cancer who respond well to induction chemotherapy and subsequently complete total neoadjuvant therapy in order to observe the organ preservation rate after total neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
1-year organ preservation rate | 1 year after completion of neoadjuvant radiotherapy
  defined as the proportion of the following two groups among the total study population：① Patients evaluated as having a clinical complete response (cCR) or near cCR at 8 weeks after radiotherapy who choose a watch-and-wait strategy and maintain cCR for 1 year; ② Patients evaluated as having a cCR or near cCR at 8 weeks after radiotherapy who ultimately undergo local excision and remain recurrence-free for 1 year without requiring salvage surgery.

SECONDARY OUTCOMES:
1-year metastasis-free survival | 1 year after total neoadjuvant therapy
  time from the start of neoadjuvant chemotherapy to the occurrence of distant metastasis
1-year overall survival | 1 year after total neoadjuvant therapy
  time from the start of neoadjuvant chemotherapy to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers are encouraged to apply for the full study protocol, study data, and analytic code upon reasonable request by contacting the primary investigator (Ziqiang Wang).
Supporting Information: Study Protocol, SAP, ICF